CLINICAL TRIAL: NCT04569773
Title: Preservation of Ovaries in Endometrial Malignancies: GYN POEM Trial
Brief Title: Choosing Ovarian Preservation or Removal Before Surgery for Endometrial Cancer
Status: Active, not recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 20-429
Record Dates: First submitted 2020-09-24; First posted 2020-09-30 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Endometrial Cancer
Keywords: Endometrial Cancer; Ovarian Preservation; Ovarian Removal; Endometrial Malignancies; GYN POEM Trial; 20-429; Memorial Sloan Kettering Cancer Center
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants undergoing surgery for clinical: Participants will be undergoing surgery for clinical stage I endometrioid endometrial cancer
  Interventions: Behavioral: Impact of Event Scale-Revised; Behavioral: Reproductive Concerns Scale; Behavioral: Decision Regret Scale

INTERVENTIONS:
Behavioral: Impact of Event Scale-Revised — The IES-R is a validated 22-item self-report scale measuring psychological stress reactions after a major life or traumatic event.1-3Items are rated with reference to the past 7 days on a 5-point scale, ranging from 0 to 4. Three subscale scores are calculated by taking the mean of the item responses: Intrustion (8 items), Avoidance (8 items), and Hyperarousal (6 items). The total score is similarly computed by taking the mean of all 22 items. All scores range from 0 to 4, with higher scores indicating higher event-related distress. Internal consistency estimates(Cronbach's alpha) for all scores range between 0.79 to 0.92.
  Other Names: IES-R
Behavioral: Reproductive Concerns Scale — The RCS is a 14-item, 5-point Likert-type self-report measure that assesses concern among cancer survivors whose reproductive ability may have been impaired or lost due to disease and/or treatment. Answers are rated on a 5-point scale (0 to 4), and a single total score is produced by summing responses to all 14 items (range, 0-56 points). A higher score represents more reproductive concerns, and a lower score represents fewer reproductive concerns. In the RCS validation study, internal consistency reliability was 0.91 among long-term female cancer survivors and 0.81 among control women.
  Other Names: RCS
Behavioral: Decision Regret Scale — The DRS is a 5-item, 5-point Likert-type self-report measure that assesses distress or remorse after a health-care decision.5 Items are rated on a scale from 1 ("strongly agree") to 5 ("strongly disagree"). Two of the statements (items 2 and 4) are phrased in the negative direction.
  A single, total score is produced by first reversing the scores of the 2 negatively phrased items, then taking the mean of the 5 items. This mean is then rescaled to range from 0 to 100 by subtracting 1, then multiplying by 25. A score of 0 indicates no regret, whereas a score of 100 indicates high regret. Internal consistency reliability coefficients for the DRS range from 0.81 to 0.92.
  Other Names: DRS

SUMMARY:
The purpose of this study is to learn more about the factors that influence decision-making before surgery (distress about cancer and/or reproductive concerns) and the possibility of regret after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Women aged ≥ 18 and ≤ 50 years
* Premenopausal
* Endometrioid histological diagnosis
* Scheduled for surgical intervention at MSKCC
* FIGO grade 1-2, clinical stage I
* Disease confined to uterus, no clear evidence of deep (≥50%) myoinvasion on imaging (MRI preferred, ultrasound optional)
* Normal ovaries on preoperative imaging
* Able to provide informed consent
* English-speaking

Exclusion Criteria:

* Known Lynch syndrome
* Prior bilateral oophorectomy
* Personal history of hormone receptor-positive breast carcinoma
* Increased risk of ovarian cancer identified on the basis of family or personal history
* Women currently on hormonal contraception, letrozole, or tamoxifen may not opt-in to AMH
* Women who recently underwent ovarian stimulation within the past 3 months may not opt-in to AMH
* Women who have pituitary dysfunction (or any pituitary disorders) may not opt-in to AMH
* Women who completed chemotherapy within <12 months may not opt-in to AMH

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients will be recruited from the Gynecology Service, Department of Surgery, at MSK. All women undergoing surgery for endometrial cancer without clear preoperative suspicion for advanced-stage disease will be screened for participation in this study. No selectivity will be exercised by the investigators to minimize bias. The specific type of surgery for each patient, as well as its timing, will be determined by the treating gynecological surgeon.
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2020-09-23 (Actual); Primary Completion 2026-09-23 (Estimated); Study Completion 2026-09-23 (Estimated)

PRIMARY OUTCOMES:
Examine the decision-making process of patients who choose to undergo or not undergo ovarian-sparing surgical treatment of endometrial cancer | Up to 12 months post-operatively
  Examine the decision-making process of patients who choose to undergo or not undergo ovarian-sparing surgical treatment of endometrial cancer to identify influencing factors-in particular, cancer-related psychological distress and reproductive concerns-and any potential decisional regrets following surgical intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Mueller, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (8):
- United States (8):
  - Hartford Healthcare (Data Collection), Hartford, Connecticut
  - Memorial Sloan Kettering Basking Ridge (All Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (All protocol activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (All protocol activities), Montvale, New Jersey
  - Memorial Sloan Kettering Cancer Center @ Suffolk (All protocol activities), Commack, New York
  - Memorial Sloan Kettering Westchester (All protocol activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Study Activities), New York, New York
  - Memorial Sloan Kettering Nassau (All protocol activities), Rockville Centre, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org